CLINICAL TRIAL: NCT06400043
Title: The Influence of an Interceptive Task on Gait in Children With Developmental Coordination Disorder Compared to Typically Developing Children
Brief Title: Dual-tasking Effect on Gait in Children With Developmental Coordination Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ONZ-2023-0650
Record Dates: First submitted 2024-05-01; First posted 2024-05-06 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Gait
Keywords: Gait analysis; Dual-tasking; EMG; Kinematics; Kinetics; Selective motor control; Developmental Coordination Disorder; DCD
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treadmill walking (Experimental): Participants will be asked to walk at different gait velocities for 1 minute. The treadmill speed will be increased incrementally at 0.1m/s intervals until just before running. The comfortable walking speed will be determined.
  Interventions: Other: Cognitive dual-task; Other: Motor dual-task

INTERVENTIONS:
Other: Cognitive dual-task — Participants will be asked to walk at comfortable walking speed while playing an additional cognitive task, namely the Stroop Color and Word Test.
Other: Motor dual-task — Participants will be asked to walk at comfortable walking speed while playing an additional motor task, namely a game that requires arm swing to hit the targets.

SUMMARY:
The aim of the study is to collect data in children with developmental coordination disorder (DCD) aged between 7 and 17 years for analyses of the gait pattern while walking at the Gait Real-time Analysis Interactive Lab (GRAIL) at the university hospital of Ghent.

Children with DCD will be asked to take a motor test (M-ABC-2) as well as walk on the treadmill during a single session of approximately 3 hours.

The following data will be collected on the GRAIL while subjects walk at different gait speeds: 3D kinematics, kinetics, and EMG.

Additionally, 3D kinematics, kinetics, and EMG data will be collected when performing either a cognitive (Stroop Color and Word Test) or motor (requiring arm swing) dual-task while walking at comfortable walking speed..

DETAILED DESCRIPTION:
The aim of the study is to collect data in children with developmental coordination disorder (DCD) aged between 7 and 17 years for analyses of the gait pattern while walking at the Gait Real-time Analysis Interactive Lab (GRAIL). This is a treadmill linked to a virtual environment used to analyse and train gait at the Children's Rehabilitation Centre of Ghent University Hospital. The data from children with DCD will be compared with typically developing children. In this study, only children with DCD will be included and the data resulting from this study will be compared to the data from the previous study in typically developing children (ID: B670201942108).

Children with DCD will be asked to take a motor test (M-ABC-2) as well as walk on the treadmill during a single session of approximately 3 hours. While walking at comfortable walking speed, two short games will be played i.e. dual-tasking. This involves both a cognitive (Stroop Colour-Word Test) and a motor (requires the use of the arms) dual task projected in the virtual environment of the GRAIL. The cognitive and motor task will be performed both while standing still (single tasking: ST) and while walking (dual tasking: DT). Simultaneously, kinetics, kinematics, and EMG data will be collected for 3D gait analysis. Using muscle synergy analysis (based on EMG data), the degree of gait automatization will be analysed. The data from children with DCD will be compared with typically developing children to determine whether a reduced gait automatization can be observed in children with DCD.

Parents will be asked to complete a screening list (CVO/DCD-Q) for motor problems in daily life. This aims as a support to the motor test (M-ABC-2), together providing additional insight into children's motor functioning (in daily life).

ELIGIBILITY:
Inclusion Criteria:

* They have an official DCD diagnosis;
* Are aged between 7 and 17 years old;
* Can walk at least 15 minutes consecutively;
* Have good or corrected vision.

Exclusion Criteria:

* They suffer from a neurological disorder;
* Take medications that affect gait and balance;
* Have undergone surgical procedures on the lower limbs in the past;
* Experience pain in their lower limbs or back at the time of testing.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Kinematics | Single point assessment, day 1
  3D kinematics of lower and upper limb joints while walking (degrees)
Kinetics | Single point assessment, day 1
  3D kinetics of lower limb joints while walking (Nm)
EMG | Single point assessment, day 1
  Muscle activity of 16 lower limb muscles (microvolts)
Muscle synergies | Single point assessment, day 1
  Synergy analysis will be conducted using the EMG data (variance accounted for -VAF)
Spatiotemporal parameters | Single point assessment, day 1
  Spatial parameters (m), temporal parameters (s), walking velocity (m/s)

SECONDARY OUTCOMES:
Gait deviation index | Single point assessment, day 1
  Based on kinematics, the lower-limb gait deviations will be calculated (degrees)
Game result (cognitive task) | Single point assessment, day 1
  Score (% correct)
Game result (motor task) | Single point assessment, day 1
  Score (% correct)

OTHER OUTCOMES:
Demographic data | Single point baseline assessment
  Gender, age
Anthropometric data (height) | Single point baseline assessment
  Height and segment lengths (cm)
Anthropometric data (weight) | Single point baseline assessment
  Weight (kg)
M-ABC-2 | Single point baseline assessment
  Standardized tool to identify motor functioning in children (standard score between 1 and 19)
  Standard scores indicate:
  * Significant motor difficulty: standard score < 6
  * Minor motor difficulties: standard score 6 or 7
  * No motor difficulty: standard score > 7
Developmental Coordination Disorder Questionnaire (DCDQ) | Single point baseline assessment
  Brief parent questionnaire to screen for coordination disorders in children (total score between 15-75)
  Children score suspected/an indication for DCD when:
  * Age 5-7: score of <47
  * Age 8-9: score of <56
  * Age 10-15: score of <58

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Bar-On, Principal Investigator — University Ghent
Locations (2):
- Belgium (2):
  - Ghent University, Ghent, East-Flanders
  - Ghent University, Ghent

IPD SHARING:
Plan to Share IPD: No